CLINICAL TRIAL: NCT04267497
Title: Phase I, Prospective, Randomised, Controlled Study on the Safety and Efficacy of Nebulised Liposomal Amphotericin as an Adjuvant Treatment for Invasive Pulmonary Aspergillosis
Brief Title: Nebulised Liposomal Amphotericin for Invasive Pulmonary Aspergillosis (NAIFI01 Study)
Acronym: NAIFI01
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Fundacion para la Investigacion Biomedica del Hospital Universitario Ramon y Cajal (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FundacionRamonCajal
Record Dates: First submitted 2019-12-24; First posted 2020-02-13 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2021-01

CONDITIONS: Invasive Pulmonary Aspergillosis
MeSH Terms: conditions — Invasive Pulmonary Aspergillosis | interventions — Amphotericin B; liposomal amphotericin B

STUDY DESIGN:
Intervention Model Description: Phase I, One-center, Prospective, Randomized and controlled study
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Nebulized Amphotericin B (Experimental): Amphotericin B.
  Interventions: Drug: Amphotericin B Liposomal 50 MG
- Nebulized Placebo (Placebo Comparator): Sterile water for injection.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Amphotericin B Liposomal 50 MG — Amphotericin B 50 mg powder for infusion diluted in 12 ml of sterile water. It will be administered by nebulized route 25 mg (6 ml), 3 times a week, for 6 weeks.
  Other Names: Ambisome
  Arms: Nebulized Amphotericin B
Other: Placebo — Sterile water for injection. It will be administered by nebulized route: 6 ml, 3 times a week for 6 weeks.
  Arms: Nebulized Placebo

SUMMARY:
The investigators aim to assess the safety and efficacy of nebulized liposomal amphotericin B (ALN) as a complementary therapy to the usual systemic treatment in patients with invasive pulmonary aspergillosis and the utility of a non-routine test as a surrogate marker of efficacy. To this end, a 3-year phase I, prospective, randomized and controlled clinical trial will be carried out in a single center, in patients with proven or probable pulmonary aspergillosis receiving routine systemic treatment. Participants will be randomized ( 1: 1) to receive ALN, 25 mg or nebulizer injection water 3 times a week, for 6 weeks. The primary objective is the safety of ALN in this scenario, including clinical tolerance and pharmacokinetic studies. Secondary objectives are presented as: a) clinical efficacy, using the following criteria: complete response, partial response, stability and progression or death, on week 12; b) microbiological efficacy, using culture, galactomannan, BDGlucan and Aspergillus PCR in induced sputum on week +6; and c) to explore the utility of the SUV ("standardized uptake value") index in PET-CT performed on week +6 in relation to a baseline PET-CT as a surrogate marker of response. The administration of ALN and placebo will be carried out by eFlowR vibrating membrane electronic nebulizers. To carry out the study, the following visits will be made: baseline, week 1,2,3,4,5,6 (efficacy and safety evaluation), 9 and 12 (overall evaluation).

DETAILED DESCRIPTION:
Phase of the clinical trial Phase I trial (pilot study), prospective, randomised, controlled trial using a drug under conditions of use not approved for the form of administration.

It is a Phase I study since the primary objective includes tolerance analysis, safety and pharmacokinetic and distribution studies of nebulized amphotericin, but when administered to patients it also carries out the preliminary assessment of the safety and efficacy of the treatment.

Primary and secondary variables

Primary variable:

Reduction of >20% of post-nebulized FVC and FEV1 in relation to values obtained before nebulization.

In each visit made during the nebulized therapy period (week 1 visit in view of week 6) the following parameters will be objectified: before and after nebulization:

* forced vital capacity (FVC)
* forced expiration volume in 1 second (FEV1) Both parameters will be measured with the Micro Spirometer; Micro Medical Ltd; Rochester UK). Repeat 3 times and obtain the higher value

Secondary variables:

* Related to tolerability and safety
* At systemic level: Fr Resp/min: Breathing rate per minute, Fr Card/min: Heart rate per minute, BP (mmHg): Systolic and diastolic blood pressure, Sat 02 (%): Percentage of oxygen saturation (digital pulse oximetry), blood test disturbances.
* At the pulmonary level: symptomatic cough, bronchospasm (auscultation), dyspnea or shortness of breath, need for bronchodilator treatment.
* Others: bad taste in mouth, nausea, dysphagia Given the practical absence of systemic passage of nebulized Ambisome confirmed in other studies, the practical absence of reported systemic reactions and given the high number of systemic events that these patients develop in relation to their underlying pathology and the use of other systemic treatments, adverse events of an extrapulmonary or systemic nature that are not considered adverse reactions (related to nebulized therapy, the object of the study) will not be collected for the study.
* related to pharmacokinetics
* Concentration of amphotericin in bronchoalveolar lavage
* Plasma amphotericin concentration Related to Effectiveness
* Radiological efficacy (including PET-CT control): Image response and PET-CT performance: Quantification of SUV metabolic uptake index in a combined positron emission tomography (PET-CT).
* Microbiological efficacy in BAL: Microbiological response in bronchoalveolar lavage (BAL): Comparison of results of calcofluor staining, fungal culture, galactomannan, BDGlucan and Aspergillus PCR of BAL samples obtained by fibrobronchoscopy
* Serum microbiological response: Comparison of results for galactomannan and BDGlucan in serum during the weeks of study follow-up

ELIGIBILITY:
Inclusion Criteria:

* Those over 18 years of age, signed by the IC or its representative, with a compatible respiratory clinic and meeting the following criteria will be included in the study: aspergillosis confirmed in sterile sample culture (e.g. lung biopsy) or with histological evidence of invasion, regardless of the patient's condition (proven aspergillosis).
* In the absence of proven aspergillosis, patients who meet all 3 conditions below are considered likely and also eligible for inclusion:

  * Clinical criteria: neutropenia (<500 neutrophils /ul), haematological malignancy, haematopoietic parent transplantation, solid organ transplantation, prolonged use of steroids, solid tumour, HIV infection, systemic diseases requiring immunosuppressive therapy, chronic obstructive pulmonary disease, cirrhosis, malnutrition, post-operative cardiac surgery or respiratory distress secondary to influenza;
  * Radiological criteria (TAC): infiltrates with halo effect, aerial meniscus, nodular, cavitated, ground glass, tree in bud or in general the presence of abnormal or persistent images refractory to antibiotherapy;
  * Microbiological criterion: isolation of Aspergillus spp in respiratory samples (whether or not associated with hyphae vision in staining techniques) or the positivity of galactomannan in serum (>0.5 x2 or >0.8 x1) or galactomannan in BAL (>1.0);

Exclusion Criteria:

* Inability or refusal of the patient (or his/her legal representative) to grant the IC.
* Pregnancy or planning to become pregnant during the course of the study. Breastfeeding.
* Formal contraindication for the administration of nebulized drugs, hypersensitivity to amphotericin.
* Patients admitted to the ICU and patients who at the time of randomization are intubated or require imminent intubation cannot be included because some studies have confirmed that nebulized Ambisome can precipitate in the breathing tubes.
* Participation in another clinical trial in the previous month or life expectancy < 1 week.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2019-10-18 (Actual); Primary Completion 2022-11-10 (Actual); Study Completion 2022-11-10 (Actual)

PRIMARY OUTCOMES:
Reduction of >20% of FVC postnebulization compared to values before amphotericin nebulization | During amphotericin treatment: week 1 to week 6
  FVC will be measured with the Micro Spirometer (Micro Medical Ltd; Rochester UK) 3 times before and after nebulization and the higher value will be recorded.
Reduction of >20% of FEV1 postnebulization compared to values before amphotericin nebulization | During amphotericin treatment: week 1 to week 6
  FEV1 will be measured with the Micro Spirometer (Micro Medical Ltd; Rochester UK) 3 times before and after nebulization and the higher value will be recorded.

SECONDARY OUTCOMES:
Fr Resp/min (Breathing rate per minute) | During amphotericin treatment: week 1 to week 6
  Change in Fr Resp/min values postnebulization compared to values before nebulization
Sat 02 (%) (Percentage of oxygen saturation) | During amphotericin treatment: week 1 to week 6
  Change in Sat 02 (%) values postnebulization compared to values before nebulization
Fr Card/min (Heart rate per minute) | During amphotericin treatment: week 1 to week 6
  Change in Card/min values postnebulization compared to values before nebulization
Number of events observed at pulmonary level. | During amphotericin treatment: week 1 to week 6
  Symptomatic cough, bronchospasm (auscultation), dyspnea or shortness of breath, need for bronchodilator treatment.
Pharmacokinetics. Concentrations of amphotericin | Week 6
  Amphotericin concentrations in bronchoalveolar lavage and in plasma.
Radiological response | Week 6
  Evaluated by PET-TC
Microbiological response. | Week 6
  Evaluated in bronchoalveolar lavage (BAL)

CONTACTS AND LOCATIONS:
Overall Officials: Sonsoles Sancho, Study Chair — President of CEIC Hospital Ramon y Cajal
Locations (1):
- Jesus Fortun, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Yes
Identifiing candidates prospectively according inclusion and exclusion criteria
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be available whiting 6 month of study completion